CLINICAL TRIAL: NCT03589963
Title: Effectiveness and Feasibility of Providing Postnatal Breastfeeding Support to Vulnerable Mothers as an Extension to the Canada Prenatal Nutrition Program
Brief Title: Providing Postnatal Breastfeeding Support Through the Canada Prenatal Nutrition Program
Acronym: PINSTEP-4
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Institutional ORE decision to stop community based research in response to COVID emergency and need to socially distance
Sponsor: University of Toronto (Other)
Collaborators: Sprott Foundation (Unknown); Parkdale Queen West Community Health Centre (Unknown)
Responsible Party: Principal Investigator, Daniel Sellen, Professor, University of Toronto
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 123345
Record Dates: First submitted 2018-07-06; First posted 2018-07-18 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Breastfeeding; Breastfeeding, Exclusive; Infant Nutrition; Complementary Feeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-intervention (No Intervention): regular CPNP programming
- Post-intervention (Experimental): regular CPNP programming plus access to postnatal lactation support
  Interventions: Behavioral: Postnatal Lactation Support

INTERVENTIONS:
Behavioral: Postnatal Lactation Support — In-home breastfeeding support delivered by professional lactation consultants and provision of a high-quality breast pump
  Arms: Post-intervention

SUMMARY:
The Canada Prenatal Nutrition Program (CPNP) aims to improve birth outcomes among Canadian women in challenging life circumstances, including those who are adolescents, newcomers, low-income or single mothers. The CPNP strongly promotes breastfeeding prenatally, resulting in high initiation rates, but continued postnatal support is needed to optimize breastfeeding duration and exclusivity.

The aim of this research is to investigate the effects of adding postnatal lactation support as an extension to the CPNP on breastfeeding duration and exclusivity in the first six months postpartum. The research will be conducted at two CPNP sites in Toronto, Parkdale Queen West Community Health Centre and The Stop Community Food Centre. A quasi-experimental design will be used to compare the infant feeding practices of CPNP clients before and after introduction of a postnatal lactation support intervention which will include in-home professional lactation support and provision of high-quality breast pumps. These services will be delivered as CPNP program components and will be accessible to all clients at the two participating sites during the post-intervention period. Infant feeding practices will be assessed by a questionnaire administered at 2 weeks, 1, 2, 3, 4, 5 and 6 months postpartum. The hypothesis is that significantly more mothers in the post-intervention group will be exclusively breastfeeding at four months postpartum. The effect is expected to be mediated through increased breastfeeding self-efficacy, which will be assessed using validated scales prenatally and at 2 weeks and 2 months postpartum.

ELIGIBILITY:
Inclusion Criteria:

* CPNP clients registered prenatally
* intention to initiate breastfeeding
* intention to remain in Toronto with the infant for 6 months postpartum
* willing to share contact information
* birth at 34 weeks gestation or later

Exclusion Criteria:

* preterm birth (below 34 weeks)
* infant has congenital abnormality or medical condition affecting feeding
* mother or infant still in hospital at 2 weeks postpartum

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 151 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2021-07-13 (Actual)

PRIMARY OUTCOMES:
Exclusive breastfeeding at 4 months postpartum | birth to 4 months postpartum
  Reported exclusive breastfeeding at four months postpartum assessed by a prospective infant feeding questionnaire

SECONDARY OUTCOMES:
Duration of any breastfeeding in the first six months postpartum | birth to 6 months postpartum
  Duration of any breastfeeding from birth to 6 months assessed by a prospective infant feeding questionnaire
Duration of exclusive breastfeeding in the first six months postpartum | birth to 6 months postpartum
  Duration of exclusive breastfeeding from birth to 6 months assessed by a prospective infant feeding questionnaire
Age of introduction of breastmilk substitutes | birth to 6 months postpartum
  Reported timing of the introduction of breastmilk substitutes from birth to 6 months in response to a prospective infant feeding questionnaire
Age of introduction of complementary foods | birth to 6 months postpartum
  Reported timing of the introduction of complementary foods from birth to 6 months in response to a prospective infant feeding questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Sellen, PhD, Principal Investigator — University of Toronto; Deborah O'Connor, PhD, Principal Investigator — University of Toronto
Locations (2):
- Canada (2):
  - Parkdale Queen West Community Health Centre, Toronto, Ontario
  - The Stop Community Food Centre, Toronto, Ontario

REFERENCES:
- [Derived] Mildon A, Francis J, Stewart S, Underhill B, Ng YM, Rousseau C, Di Ruggiero E, Dennis CL, Kiss A, O'Connor DL, Sellen DW. Associations between use of expressed human milk at 2 weeks postpartum and human milk feeding practices to 6 months: a prospective cohort study with vulnerable women in Toronto, Canada. BMJ Open. 2022 Jun 8;12(6):e055830. doi: 10.1136/bmjopen-2021-055830. PMID 35676013
- [Derived] Mildon A, Francis J, Stewart S, Underhill B, Ng YM, Rousseau C, Di Ruggiero E, Dennis CL, O'Connor DL, Sellen DW. High levels of breastmilk feeding despite a low rate of exclusive breastfeeding for 6 months in a cohort of vulnerable women in Toronto, Canada. Matern Child Nutr. 2022 Jan;18(1):e13260. doi: 10.1111/mcn.13260. Epub 2021 Aug 8. PMID 34369075
- [Derived] Mildon A, Francis J, Stewart S, Underhill B, Ng YM, Richards E, Rousseau C, Di Ruggiero E, Dennis CL, O'Connor DL, Sellen DW. Effect on breastfeeding practices of providing in-home lactation support to vulnerable women through the Canada Prenatal Nutrition Program: protocol for a pre/post intervention study. Int Breastfeed J. 2021 Jul 2;16(1):49. doi: 10.1186/s13006-021-00396-y. PMID 34215288